

## STATISTICAL ANALYSIS PLAN

# A Phase 2a Open-Label, Multi-Center Study to Evaluate the Safety and Tolerability of Multiple Doses of AT-1501 in Adults with ALS

Sponsor: Anelixis Therapeutics, LLC.

Protocol Number: AT-1501-A201

Author:

Date: 30SEP2021

Version: 1.0



# A Phase 2a Open-Label, Multi-Center Study to Evaluate the Safety and Tolerability of Multiple Doses of AT-1501 in Adults with ALS

Protocol Number: AT-1501-A201

SAP Version: 1.0

SAP Date: 30SEP2021





## **Table of Contents**

| 1. | Introduction | 6 |
|-----|--------------------------------------------------|----|
| 2. | Study Objectives | 6 |
| 2.1 | Study Endpoints | 6 |
| 2.2 | Primary Endpoint | 6 |
| 2.3 | B Exploratory Endpoints | 6 |
| 3. | Study Design and Procedures | 7 |
| 3.1 | General Study Design | 7 |
| 3.2 | 2 Schedule of Visits and Assessments | 7 |
| 4. | Study Treatments | 8 |
| 4.1 | Method of Assigning Subjects to Treatment Groups | 8 |
| 4.2 | 2 Blinding and Unblinding | 9 |
| 5. | Sample Size and Power Considerations | 9 |
| 6. | Data Preparation | 9 |
| 6.1 | I Input Data | 9 |
| 6.2 | 2 Output Data | 9 |
| 7. | Analysis Populations | 10 |
| 7.1 | Safety Analysis Set | 10 |
| 7.2 | 2 Full Analysis Set | 10 |
| 7.3 | B Evaluable Analysis Set | 10 |
| 8. | General Statistical Considerations | 10 |
| 8.1 | Missing or Inconclusive Data Handling | 10 |
| 8.2 | 2 Derivation of Analysis Screening Visit | 10 |
| 8.3 | B Definition of Baseline | 10 |
| 8.4 | 1 Data Analysis Conventions | 10 |
| 8.5 | 5 Adjustment for Multiplicity | 11 |
| 9. | Disposition of Subjects | 11 |
| 10. | Demographics and Baseline Characteristics | 12 |
| 11. | Medical History and Concomitant Medications | 12 |
| 11. | .1 Medical History | 12 |
| 11. | .2 Prior and Concomitant Medications | 12 |
| 12. | Treatment Exposure | 13 |
| 13. | Safety Analyses | 13 |
| 13. | .1 Adverse Events | 13 |
| 13. | .2 Clinical Laboratory Data | 15 |
| 13. | .3 Vital Signs | 15 |
| 13. | .4 Electrocardiogram | 15 |



| 13. | .5 Columbia Suicide Severity Rating Scale | 16 |
|-----|-------------------------------------------|----|
| 15. | Interim Analyses | 18 |
| 16. | Changes from Protocol-Stated Analyses | 19 |
| 17. | Revision History | 19 |
| 18. | Tables | 19 |
| 19. | Listings | 20 |
| 20. | Figures | 21 |



## **List of Abbreviations**

| ADA | Anti-drug Antibody |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| ALS | Amyotrophic Lateral Sclerosis |
| ALSFRS-R | ALS Functional Rating Scale - Revised |
| ATC | Anatomical Therapeutic Chemical |
| BLQ | Below the Limit of Quantitation |
| BMI | Body Mass Index |
| COVID-19 | Coronavirus Disease 2019 |
| C-SSRS | Columbia Suicide Severity Rating Scale |
| CV | Coefficient of Variation |
| DMC | Data Monitoring Committee |
| EAS | Evaluable Analysis Set |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| EDC | Electronic Data Capture |
| FAS | Full Analysis Set |
| ICH | International Conference on Harmonisation |
| IL6 | Interleukin 6 |
| IP | Investigational Product |
| IV | Intravenous |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NCI-CTCAE | National Cancer Institute Common Terminology Criteria for Adverse Events |

| PT | Preferred Term |
|------|-------------------------------------------------|
| QTcF | QT Interval Corrected with Fridericia's Formula |
| RTF | Rich Text Format |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| SDC | Statistics & Data Corporation |
| SDTM | Study Data Tabulation Model |
| SOC | System Organ Class |
| SVC | Slow Vital Capacity |
| TEAE | Treatment-Emergent Adverse Event |

WHODrug

World Health Organization Drug Dictionary



#### 1. Introduction

The purpose of this statistical analysis plan (SAP) is to describe the planned analyses and reporting for protocol AT-1501-A201, Version 04 dated 08MAR2021.

This SAP is being written with due consideration of the recommendations outlined in the most recent International Conference on Harmonisation (ICH) E9 Guideline entitled Guidance for Industry: Statistical Principles for Clinical Trials and the most recent ICH E3 Guideline entitled Guidance for Industry: Structure and Content of Clinical Study Reports.

This SAP describes the data that will be analyzed and the subject characteristics, safety and tolerability, efficacy, biomarker, immunogenicity, and pharmacokinetic (PK) assessments that will be evaluated. This SAP provides details of the specific statistical methods that will be used. The statistical analysis methods presented in this document will supersede the statistical analysis methods described in the clinical protocol. If additional analyses are required to supplement the planned analyses described in this SAP, they may be completed and will be identified in the clinical study report.

#### 2. Study Objectives

The primary objective of the study is to determine the safety and tolerability of intravenous (IV) administration of multiple doses of AT-1501 (planned 1.0, 2.0, 4.0, and 8.0 mg/kg).



#### 2.1 Study Endpoints

#### 2.2 Primary Endpoint

 Safety and tolerability variables include incidence of adverse events (AEs) and changes in physical examination, vital signs, electrocardiograms (ECGs), laboratory parameters, and the Columbia Suicide Severity Rating Scale (C-SSRS).



#### 3. Study Design and Procedures

#### 3.1 General Study Design

This is a Phase 2a, multi-center, open label, multiple dose study of AT-1501, a humanized monoclonal antibody antagonist to CD40LG. Approximately 54 adults with ALS will be enrolled into the study at up to 12 ALS treatment sites in the United States and one site in Canada.

Four ascending doses of AT-1501 (1.0 mg/kg, 2.0 mg/kg, 4.0 mg/kg, and 8.0 mg/kg) will be administered as a 1-hour IV infusion to sequentially enrolling cohorts. The 1.0 mg/kg and 2.0 mg/kg cohorts will consist of 9 participants each and the 4.0 mg/kg and 8.0 mg/kg cohorts will consist of 18 participants each. The participants in each cohort will receive 6 bi-weekly (every other week) infusions of AT-1501 over an 11-week period.

This study consists of a 4-week screening period, an 11-week dosing period in which participants are dosed once every other week, and a 4-week follow-up period. On Day 1, eligible participants will receive their first 1-hour IV infusion of AT-1501 and will be observed for at least 2 hours post infusion before being released. They will return on Weeks 3, 5, 7, 9, and 11 for subsequent infusions and will remain at the clinical site for at least 2 hours for observation and assessments before being released. Participants will be called weekly between dosing visits (Weeks 2, 4, 6, 8, 10, and 12) by a member of the research team to record AEs and changes in concomitant medications. Participants will be followed for an additional 4 weeks after their last dose to monitor for safety, with an end of study clinic visit occurring at Week 15.

Each participant will be monitored for safety throughout the study. Safety will be assessed by evaluation of AEs, changes in safety laboratory parameters, physical examination including vital signs, ECGs, and the C-SSRS.

The Data Monitoring Committee (DMC) will meet following the administration of 6 doses to a minimum of 33% of participants in each cohort to review safety data and to make dose escalation recommendations to Anelixis. The meetings for Dosing Cohorts 1 and 2 will be held after 3 participants have received 6 doses, for a total of 18 doses. The meetings for Dosing Cohorts 3 and 4 will be held after 6 participants have received 6 doses, for a total of 36 doses. The Schedule of Visits and Assessments is provided in the Appendix. Full details of each assessment and other design considerations can be found in the study protocol.

#### 3.2 Schedule of Visits and Assessments

The schedule of visits and assessments is provided in the Appendix.



The planned study week (or day) will be referred to in all tables and listings to enable reviewers to understand the assessment timing without referring to the protocol visit schedule. When assessments/samples are taken at both pre-dose and post-dose on the dosing days, the assessment will be labeled as pre-dose, 2 hours, or 3 hours as scheduled along with the planned study week (or day). Table 2 shows the scheduled study visits, their planned study week, planned study day, and the acceptable visit window from Day 1, for each study visit.

**Table 2. Scheduled Study Visits** 

| Scheduled Visit | Planned Study Week | Planned Study Day | Visit Window |
|---|---|---|---|
| Visit 1 | Screening | Screening | Day -30 to -1 |
| Visit 2 | Week 1 | Day 1 | - |
| Visit 3 | Week 2 | Day 8 | +/- 2 Days |
| Visit 4 | Week 3 | Day 15 | +/- 2 Days |
| Visit 5 | Week 4 | Day 22 | +/- 2 Days |
| Visit 6 | Week 5 | Day 29 | +/- 2 Days |
| Visit 7 | Week 6 | Day 36 | +/- 2 Days |
| Visit 8 | Week 7 | Day 43 | +/- 2 Days |
| Visit 9 | Week 8 | Day 50 | +/- 2 Days |
| Visit 10 | Week 9 | Day 57 | +/- 2 Days |
| Visit 11 | Week 10 | Day 64 | +/- 2 Days |
| Visit 12 | Week 11 | Day 71 | +/- 2 Days |
| Visit 13 | Week 12 | Day 78 | +/- 2 Days |
| Visit 14 / End of Study | Week 15 | Day 101 | +/- 7 Days |

#### 4. Study Treatments

Four ascending doses of AT-1501 (1.0 mg/kg, 2.0 mg/kg, 4.0 mg/kg, and 8.0 mg/kg) will be administered as a 1-hour IV infusion to sequentially enrolling cohorts. The 1.0 mg/kg and 2.0 mg/kg cohorts will consist of 9 participants each and the 4.0 mg/kg and 8.0 mg/kg cohorts will consist of 18 participants each. The participants in each cohort will receive 6 bi-weekly (every other week) infusions of AT-1501 over an 11-week period.

#### 4.1 Method of Assigning Subjects to Treatment Groups

The potential participant who signed the informed consent form and met all the inclusion criteria and none of the exclusion criteria will be allowed to participate. Nine participants will be enrolled into each of the 1.0 mg/kg and 2.0 mg/kg cohorts and 18 participants will be enrolled into each of the 4.0 mg/kg and 8.0 mg/kg cohorts. Dose escalation decisions will be made by Anelixis with input from the DMC and Investigators. After the decision has been made to continue dosing a cohort, the next dose cohort will be allowed to start



once the last participant enrolled to the current cohort has received their first dose. The same process will be followed to move to the next dose cohort. The planned dose escalation scheme may be amended based on review of the emerging data. Additional cohorts may be added, and smaller cohort sizes may be implemented based on safety data and AT-1501 serum concentration results.

#### 4.2 Blinding and Unblinding

This study is an open label study, therefore blinding and unblinding procedures do not apply.

#### 5. Sample Size and Power Considerations

Approximately 54 adults with ALS will be enrolled into the study. All participants will receive AT-1501. The sample size for this study is not based on formal statistical computation. The number of participants by dose group has been chosen in order to examine initial safety at lower doses

The sample size may increase in order to allow for replacement of subjects who are withdrawn or withdraw prior to receiving at least 4 infusions of AT-1501.

#### 6. Data Preparation

#### 6.1 Input Data

All clinical study data will be recorded on the electronic case report forms (eCRF) using electronic data capture (EDC) system, iMedNet<sup>TM</sup> version 1.194.1. In addition, study data which is not captured directly within the EDC system but is obtained from external vendors (chemistry, hematology, coagulation, urinalysis, serology, will also be included for analysis. These data sources are described in detail in data transfer agreements developed between data management and the respective external laboratory.

Final analysis will be carried out after the following have occurred:

- Database lock has occurred, including receipt of all final versions of external vendor data, with written authorization provided by appropriate SDC and Sponsor personnel. Any changes to the database after data have been locked can only be made with the approval of the Sponsor in consultation with SDC
- Protocol deviations have been identified and status defined (major/minor deviations).
- Analysis populations have been determined.

#### 6.2 Output Data

Data from EDC and data received from external vendors will be transferred to Biostatistics and incorporated into standard formats following the Study Data Tabulation Model (SDTM). Data will then be mapped to analysis datasets using the Analysis Data Model (ADaM). Both SDTM- and ADaM-formatted data will be used to create the subject listings, while all tables and figures will be based on the ADaM-formatted data.



SDTM will follow the SDTM version 1.8 model and will be implemented using the SDTM Implementation Guide version 3.3 and the SDTM Controlled Terminology version 2020-11-06. ADaM data will follow the ADaM version 2.1 model and will be implemented using the ADaM Implementation Guide version 1.2. Both SDTM and ADaM will be validated using Pinnacle 21 version 3.1. Any discrepancies in the validation will be noted in reviewer's guides accompanying the final data transfers.

Define.xml will be created for SDTM and ADaM using the Define-XML version 2.1 model.

#### 7. Analysis Populations

#### 7.1 Safety Analysis Set

All enrolled participants who receive at least one dose of study medication will be included in Safety Analysis Set.

#### 7.2 Full Analysis Set

All enrolled participants who receive at least one dose of study medication and at least one post-baseline measurement will be included in Full Analysis Set (FAS).

#### 7.3 Evaluable Analysis Set

The Evaluable Analysis Set (EAS) will include all treated participants who have no important protocol deviations likely to seriously affect the primary outcome of the study.

#### 8. General Statistical Considerations

#### 8.1 Missing or Inconclusive Data Handling

All analyses will be based on observed data only unless otherwise specified.

#### 8.2 Derivation of Screening Visit

Subjects may be rescreened when failing initial screening or falling out of the screening window. To incorporate the results from the rescreening visit, screening will be derived as the last visit before the dosing visit on Day 1, inclusive of unscheduled assessments. This screening result will be reported in summary tables, demographic, and study drug dosing listings.

#### 8.3 Definition of Baseline

Baseline will be defined as the last available observation among scheduled or unscheduled visits prior to administration of the first dose of study medication.

#### 8.4 Data Analysis Conventions

All data analysis described in this SAP, will be performed by SDC. Statistical programming and analyses will be performed using SAS® version 9.4 or higher. Output will be provided in rich text format (RTF) for tables and portable document format (PDF) for tables, listings, and figures using landscape orientation. Unless otherwise specified, all study data will be listed and sorted by dose group, subject ID, visit/time point, and parameter as applicable. Summary tables will be presented by dose group and visit as applicable.



Summaries for continuous and ordinal variables will include the number of observations (n), arithmetic mean, standard deviation (SD), median, minimum, and maximum. Minima and maxima will be reported with the same precision as the raw values; means and medians will be presented to one additional decimal place than reported in the raw values. Standard deviations will be presented to two additional decimal places than reported in the raw values. Summaries for discrete variables will include counts and percentages. All percentages will be rounded to one decimal place (ie, XX.X%). Change from baseline will be calculated as follow-up visit minus baseline.

Any inferential statistics produced for this study will be exploratory in nature. All statistical tests will be two-sided with a significance level of 0.05 ( $\alpha = 0.05$ ) unless otherwise specified. Confidence intervals (CI) for differences between treatment groups will be two-sided at 95% confidence unless otherwise specified. All p-values will be rounded to 4 decimal places; p-values less than 0.0001 will be presented as "<0.0001"; p-values greater than 0.9999 will be presented as ">0.9999.".

#### 8.5 Adjustment for Multiplicity

Adjustments for multiplicity will not be made in this early phase study.

#### 9. Disposition of Subjects

Disposition will be presented in terms of numbers and percentage of subjects by dose group and for all subjects. Percentages will be calculated using treated subjects as the denominator unless otherwise specified.

The number of subjects who screened, screen failed, enrolled, and treated will be presented.

The number and percentages of subjects in each analysis set (Safety, Full, and Evaluable) will be presented.

The number and percentages of subjects who completed the study or discontinued from the study will be presented. The reasons for study discontinuation will include AE, death, lost to follow-up, physician decision, protocol violation, study terminated by sponsor, withdrawal of consent, and other.

The number and percentages of subjects with any protocol deviation, major deviation, and minor deviation will be presented. Major and Minor deviations will be further classified into the following sub-categories: informed consent, inclusion/exclusion or treatment assignment, test article/study drug infusion and assignment at site, improper protocol procedures at site (missed, repeated, not per protocol), site's failure to report serious SAE/AE, visit out of window (missed), visit out of window (early, late), subject's use of prohibited concomitant medication, subject's failure to follow instructions, investigator documented review and/or signature missing, inadequate source documents, other, and COVID-19 related. The percentages for each sub-category of major or minor deviation category will be based on the total number of subjects with major or minor deviations.



Subject listings including subject disposition, inclusion/exclusion criteria, and protocol deviations, will be provided.

#### 10. Demographics and Baseline Characteristics

The demographic variables including age, sex, ethnicity, race, and female subjects' childbearing potential will be summarized using Safety Analysis Set.

Age (years) will be summarized by dose group and for all subjects using continuous descriptive statistics. In addition, age will be categorized into two age groups, <65 and >=65, and summarized using counts and percentages.

Sex, race, and ethnicity will be summarized by dose group and all subjects using discrete descriptive statistics. Subjects who record more than one race will be grouped into a single category denoted as Multiple. Female childbearing potential will be summarized by counts and percentages based on the number of females in each dose group.

Other baseline characteristics, including weight and body mass index (BMI) at the Screening visit; ALSFRS-R total score at the Screening Visit and at baseline; dyspnea, orthopnea, and respiratory insufficiency ALSFRS-R sub-scores at the Screening visit and at baseline; time since ALS symptom onset (days); and time since ALS diagnosis (days), will be summarized by dose group and for all subjects using continuous descriptive statistics.

A subject listing for demographic variables along with weight and BMI at the Screening visit will be provided. Additionally, separate subject listings for ALS diagnosis at Screening and pregnancy test results for female subjects with childbearing potential will be provided.

#### 11. Medical History and Concomitant Medications

#### 11.1 Medical History

Medical history will be coded using Medical Dictionary for Regulatory Activities (MedDRA) Version 23.1. Medical history will be summarized using discrete summary statistics by dose group by system organ class (SOC) and preferred term (PT) using the Safety Analysis Set. Percentages will be based on the number of subjects in each dose group. If a subject reports the same PT multiple times within the same SOC, that PT will only be reported once within that SOC. As with the PT, if a subject reports multiple conditions within the same SOC, that SOC will only be reported once. In the summaries, SOCs and PTs within an SOC are listed in alphabetical order. On study procedures or surgeries will be coded using MedDRA 23.1 and reported with medical history.

A subject listing for medical history including procedure or surgeries will be provided.

#### 11.2 Prior and Concomitant Medications

Prior and concomitant medications will be coded using World Health Organization Drug Dictionary (WHODrug) Global (B3, March 2020) and summarized to the therapeutic drug class (Anatomical



Therapeutic Chemical [ATC] 4 classification) and preferred name. If the ATC 4 classification is not provided, the next highest classification that is provided in the coding dictionary will be used. The preferred name will be defined as the active ingredient; if the active ingredient is not provided or includes more than two ingredients (e.g., multivitamins), then the drug name will be summarized as the preferred name.

Prior medications are those medications taken before the date of the first dose of study drug. Concomitant medications are defined as those medications listed as having been taken (1) prior to initiation of study drug administration and continuing for any period of time following the first administration of study drug or (2) starting at any time following the first administration of study drug. For any medications with missing information such as unknown start and end dates and unclear status (if taken prior to the study, or if ongoing), the medications will be reported as concomitant medications. Concomitant medications will be summarized using the Safety Analysis Set. Medications will be tabulated for each dose group using discrete summary statistics. Subjects may have more than one medication per ATC class. At each level of subject summarization, a subject will be counted once if he/she reports one or more medications. Percentages will be based on the number of subjects in each dose group. In the summaries, ATC classes and preferred names within an ATC class are listed in alphabetical order.

A subject listing of prior and concomitant medication will be provided.

#### 12. Treatment Exposure

Calculated dose (mg/kg) will be derived as described below and summarized along with total dose received (mg) by dose group and visit using continuous descriptive statistics and Safety Analysis Set. Counts and percentages for the number of doses administered will be summarized by dose group.

Calculated Dose (mg/kg) = Total Dose Received (mg) / Weight (kg).

where weight is the weight at Screening. If there is a weight change of 10% or greater from the weight at Screening to a dosing visit, the weight at the dosing visit will be used.

A subject listing of the study drug dosing will be provided along with the subject weight at each dosing visit and calculated dose (mg/kg). A subject listing of the phone calls made following the dosing week will be provided as well.

#### 13. Safety Analyses

All safety analyses will be conducted using the Safety Analysis set. Safety will be summarized by dose group.

#### 13.1 Adverse Events

An AE is any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product (which does not necessarily have a causal relationship with this treatment) reported during or after having received the investigational drug/procedure. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease



temporally associated with the use of an investigational product (IP), whether or not related to the IP. Treatment-emergent adverse events (TEAEs) are defined as any event that occurs or worsens on or after the first dose of study medication. All TEAEs will be collected from the first administration of IP until completion of the final visit.

A serious adverse event (SAE) is an AE that results in any of the following outcomes: death, life-threatening, persistent, or significant disability/incapacity, prompts a hospital admission or prolongs hospitalization, congenital anomaly/birth defect, or other important medical events. All SAEs will be collected from the time of informed consent until completion of the final visit.

All AEs will be evaluated by the Investigator/designee for duration, severity, seriousness, and relationship to investigational product. In addition, the actions taken for the AE will also be documented on the eCRF. Only symptoms that increase in severity or frequency after IP administration or new symptoms of illness will be recorded as AEs in the eCRF. If the event reflects worsening symptoms, then this should be captured in the event term. Untoward medical events which occur after signature of the informed consent but before IP administration will be recorded as medical history.

Serious adverse events recorded in the eCRF which began prior to the first dose of study medication will not be included in the summary tables but will be included in the AE data listings. AEs will be coded using MedDRA Version 23.1. Severity of AEs will be assessed as Grade 1 (lowest severity) to 5 (highest severity) using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 4.03. Relationship to study drug will be categorized as Not Related, Unlikely, Possible, Probable, and Related. Related AEs will be classified as those categorized as Probable, Possible, Related; or those missing an assessment of relationship to study drug.

An overall summary will be presented that includes the number of TEAEs and the number and percentage of subjects who experienced at least one TEAE by dose group and for all subjects. This summary will also include SAEs, drug-related TEAEs, drug-related SAEs, Grade 2 or higher TEAEs, drug-related Grade 2 or higher TEAEs, TEAEs by maximum CTCAE grade, TEAEs leading to study drug withdrawal, and TEAEs leading to death.

Separate summaries will be provided for TEAEs using discrete summary statistics and presented by dose group and for all subjects by SOC and PT. If a subject reports the same PT multiple times within the same SOC, that PT will only be reported once within that SOC. If a subject reports multiple conditions within the same SOC, that SOC will only be reported once. In the summary, SOCs and PTs within each SOC will be listed in order of decreasing frequency for all subjects. The summaries include:

- All TEAEs
- Drug-related TEAEs
- SAEs



A summary of TEAEs will be provided by dose group and for all subjects by PT only. In the summary, PTs will be listed in order of decreasing frequency for all subjects. In addition, summaries of TEAEs by maximum CTCAE grade will presented using discrete summary statistics by SOC, PT, maximum grade for each dose group and all subjects. AS To count the number of subjects with any TEAEs, if a subject has multiple TEAEs coded to the same SOC, or multiple TEAEs coded to the same PT within the same SOC, the subject will be counted once under the maximum grade.

Individual subject listing will be provided for all AEs, SAEs and AEs leading to study drug withdrawal.

#### 13.2 Clinical Laboratory Data

Clinical laboratory data including chemistry, hematology, coagulation, serology, and urinalysis are collected at Screening, pre-dose on each dosing day, and at the end of study. Continuous parameters of chemistry, hematology, coagulation, and urinalysis will be summarized using continuous descriptive statistics at each scheduled visit (including a summary of baseline values) by dose group. Change from baseline to each post-baseline visit will be summarized. Serology lab data will only be presented in a listing. Box plots of laboratory data will be presented by dose group and visit.

Subject listings of all clinical laboratory results will be provided. In addition, separate subject listings of clinical laboratory abnormal results will be provided. Laboratory tests needing to be repeated for eligibility or safety that can not be sent to the central lab may be collected at the local laboratory and will be presented in a separate listing.

#### 13.3 Vital Signs

Vital signs will be obtained at Screening; on the dosing day at pre-dose, 15 minutes into the infusion, and 1- and 2- hours post-infusion; and at the end of study visit. Vital signs, including systolic blood pressure (mmHg), diastolic blood pressure (mmHg), heart rate (bpm), respiratory rate (breaths/min), and temperature (C) will be summarized with continuous descriptive statistics at each scheduled visit (including a summary of baseline values) and time point by dose group. Change from baseline to each post-baseline visit and change from pre-dose within each visit will be summarized.

A subject listing of the vital sign results will be provided.

#### 13.4 Electrocardiogram

Electrocardiograms will be obtained at Screening, post-infusion on dosing days, and at the end of study visit. Electrocardiogram parameters, including PR interval, QRS interval, RR interval, QT interval, and QTcF (QT Interval Corrected by Fridericia's Formula), will be summarized using continuous descriptive statistics by dose group at each scheduled visit. Change from baseline to each post-baseline visit will also be summarized.

A subject listing of the ECG results will be provided.



## 13.5 Columbia Suicide Severity Rating Scale

The C-SSRS will be administered at Screening, pre-dose on each dosing day, and at the end of study. The C-SSRS includes Yes/No questions and prompts for suicidal ideation and suicidal behavior.

A subject listing of the C-SSRS results will be provided.











## 15. Interim Analyses

No interim analysis is planned for this study.



## 16. Changes from Protocol-Stated Analyses

## 17. Revision History

Documentation of revision to the SAP will commence after approval of the final version 1.0.

#### 18. Tables

Tables that will be included in the topline delivery are shown in italics, boldface font.

| Table Number | Title | Population |
|---|---|---|
| Table 14.1.1 | Subject Disposition | |
| Table 14.1.2 | Subject Demographics and Baseline Characteristics | Safety Analysis Set |
| Table 14.1.3 | Medical History | Safety Analysis Set |
| Table 14.1.4 | Concomitant Medications | Safety Analysis Set |
| Table 14.1.5 | Summary of Study Drug Dosing | Safety Analysis Set |

| Table 14.3.1.1 | Summary of Treatment-Emergent Adverse Events | Safety Analysis Set |
|---|---|---|
| Table 14.3.1.2 | Treatment-Emergent Adverse Events by System Organ Class and Preferred Term | Safety Analysis Set |
| Table 14.3.1.3 | Drug-Related Treatment-Emergent Adverse Events by<br>System Organ Class and Preferred Term | Safety Analysis Set |
| Table 14.3.1.4 | Serious Adverse Events (SAEs) by System Organ Class<br>and Preferred Term | Safety Analysis Set |
| Table 14.3.1.5 | Treatment-Emergent Adverse Events by Preferred Term | Safety Analysis Set |
| Table 14.3.1.6 | Treatment-Emergent Adverse Events by System Organ Class,<br>Preferred Term, and Maximum CTCAE Grade | Safety Analysis Set |
| Table 14.3.2.1 | Clinical Laboratory - Chemistry by Visit | Safety Analysis Set |
| Table 14.3.2.2 | Clinical Laboratory - Hematology and Coagulation by Visit | Safety Analysis Set |
| Table 14.3.2.3 | Clinical Laboratory - Urinalysis by Visit | Safety Analysis Set |
| Table 14.3.3 | Vital Signs by Visit | Safety Analysis Set |
| Table 14.3.4 | Electrocardiogram by Visit | Safety Analysis Set |



## 19. Listings

| Listing Number | Title |
|---|---|
| Listing 16.2.1 | Subject Disposition |
| Listing 16.2.2 | Inclusion/Exclusion Criteria for Screen Failed Subjects |
| Listing 16.2.3 | Protocol Deviations |
| Listing 16.2.4.1 | Demographics |
| Listing 16.2.4.2 | Pregnancy Test for Female Subjects with Childbearing Potential |
| Listing 16.2.4.3 | ALS Diagnosis |
| Listing 16.2.4.4 | Medical History |
| Listing 16.2.4.5 | Prior and Concomitant Medications |
| Listing 16.2.5.1 | Study Drug Dosing |
| Listing 16.2.5.2 | Phone Call |

| Listing 16.2.7.1 | Adverse Events |
|---|---|
| Listing 16.2.7.2 | Serious Adverse Events |
| Listing 16.2.7.3 | Adverse Events Leading to Drug Withdrawal |
| Listing 16.2.8.1.1 | Clinical Laboratory – Chemistry |
| Listing 16.2.8.1.2 | Clinical Laboratory – Hematology and Coagulation |
| Listing 16.2.8.1.3 | Clinical Laboratory – Urinalysis |
| Listing 16.2.8.1.4 | Clinical Laboratory – Serology |
| Listing 16.2.8.2.1 | Clinical Laboratory Abnormalities – Chemistry |
| Listing 16.2.8.2.2 | Clinical Laboratory Abnormalities – Hematology and Coagulation |
| Listing 16.2.8.2.3 | Clinical Laboratory Abnormalities – Urinalysis |
| Listing 16.2.8.3 | Local Clinical Laboratory Results |
| Listing 16.2.8.4 | Vital Signs |
| Listing 16.2.8.5 | Electrocardiogram |



| Listing 16.2.8.6 | Columbia Suicide Severity Rating Scale |
|------------------|----------------------------------------|
|------------------|----------------------------------------|

## 20. Figures

| Figure Number | Title | Population |
|---|---|---|
| Figure 14.2.3.1 | Box Plots of Blood Chemistry by Dose Group and Visit Safety | Safety Analysis Set |
| | Analysis Set | |
| Figure 14.2.3.2 | Box Plots of Hematology and Coagulation by Dose Group and Visit | Safety Analysis Set |
| | Safety Analysis Set | |
| Figure 14.2.3.3 | Box Plots of Urinalysis by Dose Group and Visit Safety Analysis | Safety Analysis Set |
| | Set | |
| | I . | |



Appendix: Schedule of Events

| | Screening | | Dosing | | Telephone Check | Dosing | Follow-up |
|---|---|---|---|---|---|---|---|
| Visit | 1 | | 2 | | 3, 5, 7, 9, 11, 13 | 4, 6, 8, 10, 12 | 14 |
| Study Week | Weeks -4 to - | | Week 1 | | Weeks 2, 4, 6, 8, 10<br>and 12 | Weeks 3, 5, 7, 9 and<br>11 | Week 15 |
| Study Day | Day -30 to -1 | Day 1<br>Pre-dose | Day 1<br>Dose | Day 1<br>Post-<br>dose | Days 8, 22, 36, 50,<br>64, 78<br>(+/-2 days) | Days 15, 29, 43, 57, 71<br>(+/-2 days) | Day 101<br>(+/-7days) |
| Informed Consent | X | | | | | | |
| Medical History and Demographics | X | | | | | | |
| Record Concomitant Medications | X | X | X | X | X | X | X |
| Review Eligibility Criteria | X | X | | | | | |
| Physical Examination <sup>1</sup> | X | X | | | | X | X |
| Vital Signs <sup>2</sup> | X | X | X | X | | X | X |
| Weight <sup>3</sup> | X | | | | | X | |
| Height | X | | 1 | | | | |
| ECG <sup>4</sup> | X | | | X <sup>4</sup> | | X <sup>4</sup> | X |
| COVID-19 testing <sup>14</sup> | X | | | | | | |
| Blood/Urine Samples for<br>Eligibility/Safety Testing <sup>5, 6, 7</sup> | X <sup>5</sup> | X <sup>6,7</sup> | | | | X <sup>6,7</sup> | X <sup>6</sup> |

| Spirometry <sup>12</sup> | x | X | | | | Weeks 5, 9, 11 (pre-<br>dose) | X |
|---|---|---|---|---|---|---|---|
| Colombia Suicide<br>Severity Rating Scale | х | х | | | | X (pre-dose) | X |
| AT-1501 1-hr Infusion <sup>13</sup> | | | X | | | Х | |
| Report Serious Adverse Events only | X | Х | | 12 | | | |
| Assess for All Adverse Events | | | X | X | Х | X | X |



- 1 Complete physical examination at Screening; symptom-directed physical examination at other times.
- 2 Vital signs (blood pressure, heart rate, temperature, respiration rate) are taken after being seated/supine for 5 minutes at Screening and then pre-dose, 15 minutes into the infusion and 1 and 2 hours post-infusion. Assessments performed post-infusion are timed from the end of the 1-hour infusion, not the IV-line flush. Vital signs may be collected within +5 min of the 15-minute timepoint and +15 min of the 1- and 2-hour post-infusion timepoints.
- 3 Weight for dose calculation is taken at Screening and on each dosing day pre-infusion. A weight change of 10% or greater will warrant a recalculation of the AT-1501 dose.
- 4 Post-infusion ECGs should be read on the day they are taken before the participant is released.
- 5 Eligibility testing includes serum chemistry, CBC with differential and platelet count, coagulation tests, serum pregnancy, HIV, HBC, HCV, and urinalysis
- 6 Safety testing includes serum chemistry, CBC with differential and platelet count, coagulation tests, urinalysis, and urine pregnancy test
- 7 Blood samples for safety testing pre-dose on dosing days only.
- 13 AT-1501 to be infused over 1 hour using an IV pump. Assessments performed post-infusion are timed from the end of the 1-hour infusion, not the IV-line flush.
- 14 A COVID-19 test will be conducted at Screening via nasal swab no longer than 1 week prior to their infusion. If a subject arrives at the treatment center and is symptomatic for COVID-19 subsequent testing may be administered to determine continued study eligibility.